CLINICAL TRIAL: NCT03674034
Title: A Neonatal Bimodal MR-CT Head Template
Acronym: Biomodal
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0047
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Magnetic Resonance Imaging
Keywords: MRI images; CTscan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- term: 50 CTscan and MRI images of children aged at term
  Interventions: Other: CTscan and MRI images
- one month: 50 CTscan and MRI images of children aged one month
  Interventions: Other: CTscan and MRI images
- two months: 50 CTscan and MRI images of children aged two months
  Interventions: Other: CTscan and MRI images

INTERVENTIONS:
Other: CTscan and MRI images — CTscan and MRI images segmented according to procedures previously developed by GRAMFC

SUMMARY:
This is a retrospective study based on the images contained in the database of the University Hospital of Amiens. There is no further examination. Electroencephalography (EEG) and Near-Infrared Spectroscopy (NIRS). These sources are widely used to specify the source of certain evoked potentials or to better define the sources of epileptic graphoelements, especially in the pre-surgical assessment of refractory epilepsies.

It is therefore important that these regions are more widely available in the constitution of the world, and that they are suitable for use in the design of new technologies. Although MRI is the gold standard for soft tissue segmentation, it is not suitable for bone extraction; especially in the newborn or the bone is very thin. On the other hand, CTscan is an excellent method for extracting bone. The contrast between bone and soft tissue is excellent. In this case, with the CTscan, the fontanelles are identified as discontinuities between the images of the temporal scales.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) and brain scan (CT Scan) are the two main modalities of structural brain imaging that are widely used in routine practice. The extraction of bone from MRI and CTscan images is an important step in the segmentation of the different tissues of the subjects' heads. It is indeed necessary to know precisely the electrical characteristics (conductivities) and optical (absorption, diffraction) of tissues (skin, bone, LCS, gray matter and white matter), or by electric currents or by photons. One of the major problems is the one that is not very poorly visualized in MRIs in CTscan, the bone is well individualized and that inversely the various brain structures are difficult to extract. This justifies the fact of performing a coregistration of images obtained in MRI and CTscan.

The skull of the newborn is an inhomogeneous structure. The fontanelles are invisible in MRI and identifiable in CTscan.

Electroencephalography (EEG) and Near-Infrared Spectroscopy (NIRS). These sources are widely used to specify the source of certain evoked potentials or to better define the sources of epileptic graphoelements, especially in the pre-surgical assessment of refractory epilepsies.

It is therefore important that these regions are more widely available in the constitution of the world, and that they are suitable for use in the design of new technologies.

Although MRI is the gold standard for soft tissue segmentation, it is not suitable for bone extraction; especially in the newborn or the bone is very thin. On the other hand, CTscan is an excellent method for extracting bone. The contrast between bone and soft tissue is excellent. In this case, with the CTscan, the fontanelles are identified as discontinuities between the images of the temporal scales.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 0 and 2 months new born at term
* with no structural abnormalities

Exclusion Criteria:

* infants > 2 months

Ages: 1 Day to 2 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Population 150 CTscan and MRI images of children aged between 0 and 2 months with no structural abnormalities when interpreted by the radiologist.
  An age group of 50 images of children at term, 50 images of children at one month, 50 images of children at two months for each category (MRI and CTscan) Since these images will be averaged by age group, it is not necessary to obtain the two images for each child.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
CTscan images | 2 months
  The objective of this study is to evaluate a model-based approach for extracting fontanel from CTscan images. Then, recalibrate these CT scan images in a unique repository with MRI images to obtain a composite image of different brain tissues such as brain, LCS and skin (MRI) and bone and fontanelle (CTscan).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Wallois, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No